CLINICAL TRIAL: NCT05133778
Title: The Effect of Sweet Orange and Pomegranate Extract Supplementation on Exercise Capacity: a Randomized Controlled Parallel Intervention Study in Healthy Overweight Individuals
Brief Title: The Effect of Sweet Orange and Pomegranate Extract Supplementation on Exercise Capacity in Middle-aged Adults
Acronym: Actiful2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University (Other)
Collaborators: BioActor B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Actiful2
Record Dates: First submitted 2021-10-26; First posted 2021-11-24 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Exercise Capacity
Keywords: Sweet orange; Pomegranate; Polyphenols; Exercise capacity; Ekblom-bak

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled parallel trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sweet orange and pomegranate extract (Experimental): Supplementation
  Interventions: Dietary Supplement: Sweet orange and pomegranate extract
- Maltodextrin (Placebo Comparator): Supplementation
  Interventions: Other: Maltodextrin control

INTERVENTIONS:
Dietary Supplement: Sweet orange and pomegranate extract — From the daily 650mg total supplementation of the investigational product, 250 mg will be of pomegranate extract containing 100mg of punicalagin. The remaining 400 mg will consist of sweet orange peel extract containing 360 mg of hesperidin.
  Arms: Sweet orange and pomegranate extract
Other: Maltodextrin control — Supplementation with 760 mg maltodextrin
  Arms: Maltodextrin

SUMMARY:
The aim of the present study is to investigate the effect of 12-week long daily administration of a sweet orange and pomegranate extract on exercise capacity in healthy adults.

DETAILED DESCRIPTION:
Background of the study: Polyphenols have been studied for their protective effect against the development of ROS-related diseases like cancers, cardiovascular diseases, diabetes, osteoporosis, and neurodegenerative diseases. The combined supplementation of pomegranate and sweet orange polyphenols could be an effective strategy to improve exercise performance, due to their antioxidant character and ability to stimulate NO production, to stimulate mitochondrial biogenesis and to accelerate muscle repair and decrease muscle tissue damage. The study aims to assess the effect of a combined supplementation of pomegranate and sweet orange extract on exercise capacity, physical activity, muscle strength and quality of life in healthy adults.

Objective of the study: The aim of the present study is to investigate the effect of 12-week long daily administration of a sweet orange and pomegranate extract on exercise capacity in healthy adults (40 - 65 y).

Study design: Randomized, double-blind, placebo-controlled parallel trial

Study population: Healthy, overweight, sedentary adults between 40 and 65 years old.

Intervention: 12-week supplementation with 650 mg sweet orange and pomegranate extract (2 capsules per day) compared to placebo (760 mg maltodextrin).

Primary outcome of the study: Change in aerobic capacity (VO2max), assessed with an Ekblom-Bak submaximal cycling test.

Secondary study parameters/outcome of the study:

* Daily physical activity as determined by accelerometer
* Dietary intake as measured by a 3-day food record
* Handgrip strength
* Muscle cell proliferation and differentiation and mitochondrial biogenesis assessed in skeletal muscle biopsies
* Quality of Life as measured by the WHO-QOL-100 questionnaire
* General health as measured by SF-36 questionnaire
* Vitality as measured by the Dutch Vitality Questionnaire (Vita-16)
* Cardiometabolic health biomarkers, cortisol, C-reactive protein determined with ELISA
* Antioxidative capacity measured with a Trolox equivalent antioxidant capacity (TEAC) assay

ELIGIBILITY:
Inclusion Criteria:

* Healthy male/female (based on medical history provided during a general health questionnaire)
* Age between 40 - 65 yrs
* Overweight (BMI ≥25 to ≤29.9 kg/m2)
* Sedentary subjects (Low Level [<600 MET-minutes/week] as assessed by the Physical Activity Questionnaire (IPAQ))

Exclusion Criteria:

* Allergy to test product/control or citrus fruits and pomegranate
* Medical conditions that might interfere with endpoints or compromise participant safety during testing (e.g. Cardiovascular diseases, cancer, Parkinson's disease, Gastrointestinal diseases or abdominal surgery) to be decided by the principal investigator
* Use of medication that might interfere with endpoints (i.e.: β-blockers, antioxidant, antidepressants)
* High fasting blood glucose (FBG ≥100 mg/dL)
* Recent skeletal muscle injury in less than one month before the start of the study
* Use of antibiotics within 3 months prior to Visit 2
* Use of probiotics or supplements containing vitamins, minerals or antioxidants four weeks prior to Visit 2
* Regular smoking (including use of e-cigarettes)
* Inability to correctly perform the PA test during screening/familiarization
* Abuse of alcohol (alcohol consumption >20 units/week) and/or drugs
* Plans to change diet or medication for the duration of the study
* Treatment with an investigational drug (phase 1-3) 180 days before the start of the study
* Inability to understand study information and/or communicate with staff

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Change in endurance capacity | 12 weeks
  An Ekblom-bak cycling test is used to estimate the maximal oxygen consumption

SECONDARY OUTCOMES:
Change in Daily physical activity | 12 weeks
  Measured with an accelerometer
Change in Handgrip strength | 12 weeks
  Measured with a dynamometer
Change in Self reported quality of life | 12 weeks
  Measured with the World Health Organization Quality of Life (WHO-QOL-100) questionnaire. For 6 domains (including physical, psychological, level of independence, social relationships, environment and religion/personal beliefs), a score will be calculated between 2 - 40 in which a higher score indicates better quality of life.
Change in General health | 12 weeks
  Measured with the 36-Item Short Form Health Survey. For 4 domains (including functional status, wellbeing, general health and change in health), a score will be calculated between 0 - 100 in which a higher score indicates better health.
Change in Vitality | 12 weeks
  Measured with the vita-16 questionnaire. For 4 domains (including energy, motivation, resilience and overall vitality), a score will be calculated between 1 - 7 in which a higher score indicates higher vitality.
Change in Glucose levels | 12 weeks
  Measured in blood samples
Change in Cholesterol levels | 12 weeks
  Measured in blood samples
Change in Triglyceride levels | 12 weeks
  Measured in blood samples
Change in Insulin levels | 12 weeks
  Measured in blood samples
Change in Cortisol levels | 12 weeks
  Measured in blood samples
Change in C-reactive protein levels | 12 weeks
  Measured in blood samples
Change in Antioxidative capacity | 12 weeks
  Measured with a TEAC assay in blood
Change in Cell elongation index | 12 weeks
  Measured with immunohistochemistry in muscle tissue samples
Change in Muscle proliferation (marker Pax7) | 12 weeks
  Measured with qPCR in muscle tissue samples
Change in Muscle differentiation (marker MyoD) | 12 weeks
  Measured with qPCR in muscle tissue samples
Change in Muscle differentiation (marker Myogenin) | 12 weeks
  Measured with qPCR in muscle tissue samples
Change in Muscle differentiation (marker Myosin Heavy Chain) | 12 weeks
  Measured with qPCR in muscle tissue samples
Change in Muscle mitochondrial biogenesis (marker PGC1alpha) | 12 weeks
  Measured with qPCR in muscle tissue samples
Change in Muscle metabolism (marker Glut4) | 12 weeks
  Measured with qPCR in muscle tissue samples
Change in Muscle redox biology (marker GCLC) | 12 weeks
  Measured with qPCR in muscle tissue samples
Change in Muscle redox biology (marker Hmox1) | 12 weeks
  Measured with qPCR in muscle tissue samples

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No